CLINICAL TRIAL: NCT04221347
Title: Early Diagnostics of Hepatocellular Carcinoma in Patients With Liver Cirrhosis by Novel Molecular Spectrometric Biomarkers in Blood Plasma
Brief Title: Novel Molecular Spectrometric Biomarkers in Blood Plasma as an Early Diagnostic Tool in HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Military University Hospital, Prague (Other)
Collaborators: University of Chemistry and Technology, Prague (Unknown)
Responsible Party: Principal Investigator, Petr Hribek, MD, Military University Hospital, Prague
Other Study IDs: Does not exist, not required
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma; Cirrhosis, Liver
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Liver Cirrhosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A - Hepatocellular carcinoma: Patients with with proved hepatocellular carcinoma in cirrhosis.
  N=100
  Interventions: Other: blood sampling
- Group B - Cirrhosis: Cirrhotics of multiple aethiology will be sampled for spectroscopy in order to detect possible differences among cirrhotics with and without subsequent hepatocellular carcinoma.
  N=100
  Interventions: Other: blood sampling
- Group C - Healthy controls: Healthy controls - healthy military personnel. N=50
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — blood samples will be taken in specified time points

SUMMARY:
Due to providing valuable clinical information while being minimally invasive, blood-based testing will most likely be a prerequisite for future large-scale screening of high-risk populations. As a variety of pathological processes, including carcinogenesis, may cause changes in both the concentration and the structure and spatial arrangement of body biomolecules, the spectroscopic analysis of blood-based derivatives appears to be an appropriate tool for the early detection thereof. The differences observed in the spectral response of healthy individuals and patients may also be specific to a particular type/stage of the disease and, thus, may serve as a reliable diagnostic marker. In order to find sufficiently specific and sensitive biomarkers of early stages of degenerative and cancerous diseases, the co-applicant group at the Department of Analytical Chemistry, University of Chemistry and Technology Prague (UCT Prague), developed a unique approach for the spectroscopic analysis of blood plasma. Using the highly specialized, structure-sensitive methods of chiroptical spectroscopy (electronic circular dichroism - ECD, Raman optical activity - ROA) combined with conventional infrared (IR) and Raman spectroscopy, the first pilot studies yielded promising results with respect to the identification of spectral markers for pancreatic cancer, colon cancer and type 1 diabetes mellitus. In addition, metabolomics appears to be a very progressive approach to finding potentially suitable molecules to distinguish between healthy and cancer-affected individuals. Therefore, the investigators believes that this multimodal approach will allow for the identification of hepatocellular carcinoma (HCC). In our research, the focus will be on the identification of novel biomarkers in blood plasma that would exhibit sufficient sensitivity and specificity to detect early and potentially curable HCC stages, and that would be potentially useful for routine screening of this disease in well-defined at-risk groups.

DETAILED DESCRIPTION:
Subjects: Patient recruitment will be performed at the Department of Gastroenterology, Hepatology and Metabolism at the Internal Clinic of the First Faculty of Medicine of the Charles University and the Military University Hospital in Prague (MUH Prague). The selection of sample set sizes is clarified below (subsection Data collection and statistical analysis).

Group A: ~100 patients with liver cirrhosis with the HCC diagnosis confirmed according to standard diagnostic criteria published recently by European Association for the study of the liver (EASL). Patients of all HCC stages according to Barcelona Clinic Liver Cancer (BCLC), in our department ~40-50 patients per year, will be included.

Group B: ~100 patients with liver cirrhosis without HCC or dysplastic nodules at the time of examination and within the next 12 months of follow-up. The patients will be monitored by regular clinical visits with general laboratory exams and liver ultrasound in 6-month intervals (recommended surveillance for patients with liver cirrhosis in risk of HCC development).

Group C: ~50 healthy volunteers without liver cirrhosis (Czech Army recruits, Czech Army active military personnel).

Routinely examined biochemistry (e.g. total protein, albumin, alpha feto protein, etc.) of all studied groups will be correlated with the newly identified spectroscopic/metabolomic biomarkers. A signed informed consent will be secured from each subject included in the study (Inclusion/exclusion criteria listed below). Plasma preparation: Following the already established procedure for sample collection, preparation and analysis, the whole anticoagulant-treated (K3EDTA) blood of all subjects will be collected by venipuncture and centrifuged at 1500 × g for 10 minutes. The plasma fractions will be frozen immediately (stored at -80 °C) and transported to the UCT Prague for spectroscopic and metabolomics analyses. Prior to each analysis, the samples will be thawed at room temperature (~25 °C) and centrifuged through a 0.45 μm membrane filter at 13,000 × g for 10 minutes. Subsequently, the spectral measurements will be carried out (in the case of ROA and Raman, a kinetic fluorescence quencher will be added to suppress the spectrally broad background of large amplitude, which overlaps the signals of interest and is caused by a high content of fluorescing molecules in blood plasma).

Spectroscopic analysis: To meet the project objectives, the investigators will utilize a unique combination of two chiroptical methods - ECD and ROA - supplemented by non-polarized variants - IR absorption and Raman spectroscopy. While ECD detects the absorption difference between left and right circularly polarized radiation, the commercially available scattered circular polarization ROA setup operates with the small intensity difference between the circularly polarized components in the scattered light using non-polarized incident radiation. Both of these methods exhibit inherent sensitivity to the 3D structure and conformation of several chiral biomolecules, such as peptides, proteins, saccharides, nucleic acids and others (20). Some of these types of compounds might be among those, whose 3D structure or concentration in blood plasma varies during HCC development. While ECD sensitively reflects the overall conformation of chiral molecules, ROA focuses on particular bond types; and thus, reflects rather the structural details. In addition to the peptide-backbone bands from regular secondary structure elements, specifically helices and beta-sheets, the ROA spectra contain distinct bands from loops and turns and, as such; they provide information on the tertiary structure. Therefore, the simultaneous use of ECD, ROA and the non-polarized spectroscopic methods will enhance the reliability of the particular findings.

Moreover, combining different analytical approaches and technologies not yet established in clinical practice will increase the likelihood of detecting minor changes within the spectral features reflecting the conformational and concentration alterations of the HCC-related molecules and/or their metabolites in blood plasma. To the best of our knowledge, our laboratory at the Department of Analytical Chemistry, UCT Prague is the only one in the world to have all of these techniques available, simultaneously having a long-term experience with biofluid analysis. All equipment used for the analyses is commercially available and, thus; may be purchased by clinical laboratories.

ELIGIBILITY:
Inclusion criteria:

Group A

* age 18-80 years, signed informed consent
* proved liver cirrhosis based on at least one of the following criteria: histopathological finding in liver biopsy, non-invasive procedures (transient elastography (Fibroscan by Echosens, France) and / or shear-wave elastography, evidence of portal hypertension, history of cirrhosis decompensation (variceal bleeding, jaundice, hepatic encephalopathy, ascites, edema)
* HCC confirmed by EASL diagnostic algorithm

Group B

* age 18-80 years, signed informed consent proved liver cirrhosis based on at least one of the following criteria: histopathological finding in liver biopsy, noninvasive procedures (transient elastography (Fibroscan by Echosens, France) and or shear-wave elastography), evidence of portal hypertension, history of cirrhosis decompensation (variceal bleeding, jaundice, hepatic encephalopathy, ascites, edema)
* HCC excluded according to: EASL diagnostic algorithm at baseline, negative liver ultrasound (no suspicious nodule in cirrhosis) during at least 2 examinations in 6 - month intervals (e.g. 12 months after baseline)

Group C

* age 18-65 years, signed informed consent
* approved Czech Army recruits and active military personnel after regular examinations with normal outcome (vital functions, ECG, blood count, blood biochemistry and urine tests, chest X-ray, physical examination)

Exclusion criteria:

* severe co-morbidities (i.e. advanced chronic heart failure, chronic renal insufficiency stage 4 and above, long-term poorly compensated diabetes mellitus with severe complications)
* absence of liver cirrhosis
* history of any other cancer than HCC
* pregnancy
* estimated patient non-compliance and/or not signing of the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group A: cca 100 patients with liver cirrhosis with the HCC diagnosis confirmed according to standard diagnostic criteria published recently by EASL. Patients of all HCC stages according to BCLC (in our department cca 40-50 patients per year) will be included
  Group B: cca 100 patients with liver cirrhosis without HCC or dysplastic nodules at the time of examination and within the next 12 months of follow-up. The patients will be monitored by regular clinical visits with general laboratory exams and liver ultrasound in 6-month intervals (recommended surveillance for patients with liver cirrhosis in risk of HCC development)
  Group C: cca 50 healthy volunteers without liver cirrhosis (Czech Army active military personnel)
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of spectroscopic markers differences among specified groups | 6 yrs
  The main aim is to identify potential HCC biomarkers accessible in blood by using methods of conventional molecular spectroscopy (Raman and infrared absorption) in combination with structure-sensitive chiroptical techniques (electronic circular dichroism and Raman optical activity) and a metabolomics analysis.

SECONDARY OUTCOMES:
Measure of sensitivity and specificity of identified biomarkers for diagnosis HCC | 6 yrs
  To evaluate specificity and sensitivity of the newly identified biomarkers for the early diagnosis of HCC in patients with liver cirrhosis.
Measure of sensitivity and specificity of identified biomarkers for surveillance of HCC | 6 yrs
  To investigate the potential model for the differentiation of premalignant dysplastic nodules and early HCC.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Military Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hribek P, Vrtelka O, Kralova K, Klasova J, Fouskova M, Habartova L, Kubickova K, Kupsa T, Tuma T, Setnicka V, Urbanek P. Efficacy of blood plasma spectroscopy for early liver cancer diagnostics in obese patients. Ann Hepatol. 2024 Sep-Oct;29(5):101519. doi: 10.1016/j.aohep.2024.101519. Epub 2024 Jun 10. PMID 38866366